CLINICAL TRIAL: NCT03851055
Title: Effect of Zinc Supplementation on Glucose Homeostasis in Patients With β-Thalassemia Major Complicated With Diabetes Mellitus
Brief Title: Zinc Supplementation in Patients With β-Thalassemia Major Complicated With Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nancy Samir Elbarbary, Professor of Pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ain shams Pediatrics 3082019
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Beta-thalassemia Major Complicated With Diabetes
Keywords: Zinc; blood glucose; diabetes; beta thalassemia
MeSH Terms: conditions — Diabetes Mellitus; beta-Thalassemia | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Active Comparator): will receive zinc supplementation
  Interventions: Drug: Zinc
- Control group (No Intervention): Patients will receive placebo only

INTERVENTIONS:
Drug: Zinc — One arm will receive Zinc Second arm will receive placebo
  Arms: intervention group

SUMMARY:
Beta-thalassemia represents a group of recessive inherited hemoglobin disorders characterized by reduced synthesis of β-globin chain. The homozygous state (β-thalassemia major) "TM" results in severe anemia, which needs regular blood transfusion . The life expectancy in patients with TM has increased due to therapeutically management, such as frequent transfusion, desferal administration and bone marrow transplantation. Diabetes is clinically characterized by hyperglycemia due to either low circulating concentrations of, or decreased sensitivity to, insulin. Patients with TM typically exhibit β-cell or insulin insufficiency, and may develop diabetes due to toxic levels of iron in their pancreas, one of the strongest predictors of β-cell destruction. By contrast, hyperinsulinemia, secondary to insulin resistance, with normal glucose tolerance has also been observed.

The pathogenic mechanisms leading from siderosis to diabetes are poorly understood.

DETAILED DESCRIPTION:
Zinc(Zn) is a critical trace element in human health. Zinc has a potential to be utilized for the treatment of type 2 diabetes; however, evidence suggests that the effect of Zn on type 2 diabetes remains unclear. Up to 85% of the whole body Zn content is found in muscle and bones, with 11% in the skin and liver .Zn is an indispensable co-factor for more than 300 enzymes involved in metabolism and also reportedly plays a role in aging, immune system, apoptosis, and oxidative stress.

Although the effect of zinc supplementation in the improvement of oxidative stress is controversial, one of the causes that the oxidative stress is present in patients with type 2 diabetes is the change in zinc metabolism. Recent studies have demonstrated that the islet-restricted zinc transporter, ZnT8 (SLC30A8), regulates insulin secretion and hepatic insulin clearance, suggesting that Zn is a key biological factor in glucose homeostasis and the risk of developing type 2 diabetes.

In patients without thalassemia, there is a rich body of literature focused on the "diabetogenic effects" of altered zinc status.

Zinc supplementation has even been suggested as an adjunct therapy in the management of non-thalassemia related diabetes .Functional zinc deficiency exists in a contemporary sample of healthy β-thalassemic patients. An estimated 20% to 30% of patients with β-thalassemia are zinc deficient. The high prevalence is thought to be related to a combination of increased urinary losses compounded by elevated requirements.

Glucose homeostasis and its relation to Zinc status has not been widely studied especially in Egyptian children and adolescents with β-thalassemia major.

The aim of this study is to:

1. Assess zinc status in patients with β-thalassemia major and diabetes mellitus and its relation to clinical and laboratory parameters of these patients.
2. Effect of zinc supplementation on glucose homeostasis in patients with β-thalassemia major and diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with β-thalassemia major and diabetes confirmed by history, examination and investigation.
* Patients on regular visits to clinic.
* Age more than 10 years old.

Exclusion Criteria:

* Those who refused to lay informed consent.
* Those below age limit.
* Patients with other disorders that may affect glucose homeostasis rather than TM.
* Patients with autoimmune disease, collagen diseases, infections, tumors, hematological diseases other than Thalassemia major.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose mg/dl | 12 weeks
  the change in fasting blood glucose level after the 12 weeks of treatment in the intervention group when compared to the placebo group.

SECONDARY OUTCOMES:
HbA1c% | 12 weeks
  changes in HbA1c% levels
fructosamine mg/dl | 12 weeks
  changes in fructosamine levels mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy Elbarbary, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Patients data and identity are totally anonymous to the study group

REFERENCES:
- [Background] Gamberini MR, Fortini M, De Sanctis V, Gilli G, Testa MR. Diabetes mellitus and impaired glucose tolerance in thalassaemia major: incidence, prevalence, risk factors and survival in patients followed in the Ferrara Center. Pediatr Endocrinol Rev. 2004 Dec;2 Suppl 2:285-91. PMID 16462713
- [Background] Capdor J, Foster M, Petocz P, Samman S. Zinc and glycemic control: a meta-analysis of randomised placebo controlled supplementation trials in humans. J Trace Elem Med Biol. 2013 Apr;27(2):137-42. doi: 10.1016/j.jtemb.2012.08.001. Epub 2012 Nov 6. PMID 23137858
- [Background] Fung EB, Kwiatkowski JL, Huang JN, Gildengorin G, King JC, Vichinsky EP. Zinc supplementation improves bone density in patients with thalassemia: a double-blind, randomized, placebo-controlled trial. Am J Clin Nutr. 2013 Oct;98(4):960-71. doi: 10.3945/ajcn.112.049221. Epub 2013 Aug 14. PMID 23945720